CLINICAL TRIAL: NCT05174221
Title: A Phase 1b, Multicenter, Open-Label Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Mezagitamab (TAK-079) in Patients With Primary IgA Nephropathy in Combination With Stable Background Therapy
Brief Title: A Study of Mezagitamab in Adults With Primary Immunoglobulin A Nephropathy Receiving Stable Background Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-079-1006; 2024-516743-34-00 (EU CTIS Number: EU CT Number); jRCT2011220009 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-12-14; First posted 2021-12-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Kidney Disease; Glomerulonephritis
Keywords: Drug Therapy
MeSH Terms: conditions — Kidney Diseases; Glomerulonephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mezagitamab (Experimental): Mezagitamab, subcutaneous injection, once weekly for 8 weeks then once every 2 weeks for 16 weeks in the Main Study. Same dosing regimen will be repeated in LTE Retreatment Period.
  Interventions: Drug: Mezagitamab

INTERVENTIONS:
Drug: Mezagitamab — TAK-079 subcutaneous injection.
  Other Names: TAK-079

SUMMARY:
This study will have two parts. The main aims are to:

* check the side effects from mezagitamab.
* check for long-term side effects from mezagitamab.

Before starting the study, participants will be asked to provide a 24-hour urine sample. A few weeks later, if enrolled they will begin receiving a subcutaneous injection (under the skin) of mezagitamab once a week for 8 weeks then once every 2 weeks for 16 weeks. When treatment has ended, there will be a 24-week follow-up period.

Participants who receive benefit from the treatment may continue in the second part of the study where they will be monitored for up to 96 weeks and possibly retreated for another 24 weeks.

DETAILED DESCRIPTION:
The drug being tested in this study is called mezagitamab. Mezagitamab is being tested for the first time in this patient population and might help to treat people who have Primary Immunoglobulin (IgA) Nephropathy. This study will evaluate the safety, tolerability, pharmacokinetics, and efficacy of mezagitamab in combination with stable background therapy.

The study will enroll approximately 16 participants. The study will consist of 2 key components: a main study and a long-term extension (LTE) study, which includes an observation period and a retreatment period. The observation period of the LTE study is a non-interventional study segment and the retreatment period of the LTE study consists of a redosing period in which participants will be administered mezagitamab at the same dose level as in the main study. Only participants who have a positive outcome during the main study will enter LTE study.

Participants will be enrolled to the following cohort:

• Mezagitamab

This multi-center trial will be conducted in the United States, Europe, and Asia Pacific. The overall time to participate in this study is approximately 154 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Renal biopsy report supporting diagnosis of primary IgAN or IgA vasculitis-associated nephritis within 10 years prior to the screening visit.
2. UPCR greater than or equal to (>=) 1 milligram per milligram (mg/mg) or urine protein excretion (UPE) >=1 gram per day (g/day) by 24-hour urine collection during the screening period.
3. Estimated glomerular filtration rate (eGFR) >=45 milliliter per minute per 1.73 square meter (mL/min/1.73m^2) at screening.
4. Receiving stable background therapy for IgAN (angiotensin-converting enzyme inhibitor [ACE-I] or angiotensin receptor blocker [ARB]) for 12 weeks prior to screening. The ACE-I and ARB dose should represent the maximum tolerated or maximum labeled dose, as determined by the investigator, for a minimum of 3 months and remain stable during the entire duration of the study.

Exclusion Criteria:

1. Kidney biopsy confirming significant renal disease other than IgAN.
2. Secondary IgAN (such as with significant liver disease, inflammatory bowel disease, and seronegative spondyloarthropathies).
3. Evidence of rapidly progressive glomerulonephritis (loss of >=50 percent (%) of eGFR within 3 months prior to the screening visit).
4. Diagnosis of nephrotic syndrome defined as 24-hour proteinuria greater than (>) 3.5 g/day, hypoalbuminemia (smaller than [<] 30 g/L) with or without peripheral edema at the screening visit.
5. Diagnosis of acute active extrarenal IgA vasculitis (Henoch-Schönlein purpura) manifested by the involvement of other organs (palpable purpura, abdominal pain, and arthritis) at the screening visit and within 1 year prior to the screening visit.
6. Previous treatment with immunosuppressive agents such as cyclophosphamide, mycophenolate mofetil (MMF), cyclosporine, azathioprine, calcineurin inhibitors within 6 months prior to the screening visit or expected use of any of these agents for the duration of the study.
7. Use of systemic corticosteroids within 4 months from screening visit or expected use for the duration of the study.

   Use of B-cell-directed biologic therapies such as blisibimod, belimumab, rituximab, ocrelizumab or have used other biologics (example, anti-tumor necrosis factor [TNF], abatacept, anti-interleukin [IL]-6) within 6 months prior to the screening visit or expected use of any of these agents for the duration of the study.
8. Participation in another investigational study within 4 weeks or 5 half-lives of study drug, whichever is longer, before the screening visit (the 4-week window is derived from the date of the last study procedure, and/or AE related to the study procedure in the previous study, to the screening visit of the current study) or expected use of an investigational agent from another investigational study during the time of this study.
9. Administration of any vaccine within 28 days before the screening visit or of any live or live-attenuated vaccination planned for the duration of the study.
10. An opportunistic infection smaller than or equal to (<=) 12 weeks before screening visit or currently receiving treatment for a chronic opportunistic infection, such as tuberculosis (TB), pneumocystis pneumonia, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria. A mild, localized herpes simplex infection within 12 weeks of study dosing is allowed, as long as the lesion has resolved prior to Day 1.
11. A positive T-cell interferon-gamma release assay (TIGRA) (result through QuantiFERON-TB Gold test or T-Spot/Elispot) at the screening visit.
12. A positive test result for hepatitis B surface antigen, or hepatitis B core antibody, or hepatitis C antibody, or HIV antibody/antigen at screening. However, an individual who has a known history of chronic hepatitis C and has been treated and fully cured of the disease, confirmed with a negative hepatitis C virus RNA polymerase chain reaction (PCR) test at screening, is not excluded on the basis of the positive hepatitis C antibody alone.
13. Inadequate organ and bone marrow function at screening visit.
14. Presence of uncontrolled or New York Heart Association (NYHA 1994) Class 3 or 4 congestive heart failure at the screening visit.
15. Uncontrolled diabetes manifested by glycosylated hemoglobin (HbA1c) >8% at the screening visit.
16. Current malignancy or history of malignancy during the previous 5 years, except adequately treated basal cell or squamous cell carcinomas of the skin or carcinoma in situ/cervical intraepithelial neoplasia of the uterine cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Main Study: Percentage of Participants With one or More Treatment-emergent Adverse Events (TEAEs), Grade 3 or Higher TEAEs, Serious Adverse Events (SAEs), and Adverse Events (AEs) Leading to Mezagitamab Discontinuation | Up to Week 48
  The severity of TEAEs will be graded using National cancer institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
LTE Observation Period: Percentage of Participants With one or More TEAEs, Grade 3 or Higher TEAEs and SAEs | Up to Week 96
  The severity of TEAEs will be graded using NCI-CTCAE version 5.0.
LTE Retreatment Period: Percentage of Participants With one or More TEAEs, SAEs, Grade 3 or Higher TEAEs and AEs leading to Mezagitamab Discontinuation | Retreatment Week 0 to 48
  The severity of TEAEs will be graded using NCI-CTCAE version 5.0.

SECONDARY OUTCOMES:
Main Study: Ctrough: Observed Serum Trough Concentrations of Mezagitamab | Week 0 Pre-dose and at multiple time points (up to Week 48)
Main Study: Serum IgA Levels | Week 0 Pre-dose and at multiple time points (up to Week 48)
Main Study: Percent Change From Baseline in Proteinuria Based on Urine Protein to Creatinine Ratio (UPCR) | Week 36
  UPCR is calculated by dividing the concentration of protein (milligram per deciliter [mg/dL]) in urine by the urine creatinine concentration (mg/dL).
Main Study: Percentage of Participants Based on Antidrug Antibody (ADA) Levels in Serum | Up to Week 48
  Percentage of participants in each category of the immunogenicity status (ADA-negative, ADA-positive and titer) will be determined in this study.
LTE Observation Period: Serum IgA Levels | Week 56 Pre-dose and at multiple time points (up to Week 96)
LTE Observation Period: Percent Change From Baseline in Proteinuria Based on UPCR | Up to Week 96
  UPCR is calculated by dividing the concentration of protein (mg/dL) in urine by the urine creatinine concentration (mg/dL).
LTE Observation Period: Percentage of Participants Based on ADA Levels in Serum | Up to Week 96
LTE Retreatment Period: Percentage of Participants Based on ADA Levels in Serum | Up to Retreatment Week 48
  Percentage of participants in each category of the immunogenicity status (ADA-negative, ADA-positive and titer) will be determined in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (26):
- United States (3):
  - Amicis Research Center - Northridge - Nordhoff, Northridge, California
  - Boise Kidney and Hypertension Institute - Frenova, Nampa, Idaho
  - NorthShore University HealthSystem, Evanston, Illinois
- Australia (3):
  - Core Research Group, Milton, Queensland
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- China (3):
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
- Hungary (2):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád megye
  - Semmelweis Egyetem, Budapest
- ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia, Lombardy, Italy
- Japan (4):
  - Kasugai Municipal Hospital, Kasugai-Shi, Aiti
  - Fujita Health University Hospital, Toyoake-shi, Aiti
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo City General Hospital, Sapporo, Hokkaido
- National University Hospital- Singapore, Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Ajou University Hospital, Suwon
- Spain (3):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Fundacio Puigvert, Barcelona
- Taiwan (2):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
- United Kingdom (2):
  - Leicester General Hospital, Leicester, Leicestershire
  - Hull Royal Infirmary, Hull

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/7f3e474338f74829?idFilter=%5B%22TAK-079-1006%22%5D